CLINICAL TRIAL: NCT06617780
Title: Radiological Criteria for Instability in Distal Radius Fractures
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Bergesenstiftelsen (Unknown)
Responsible Party: Principal Investigator, Lene Bergendal Solberg, Senior physician and postdoctoral fellow, Orthopedic Department, Oslo University Hospital, Oslo University Hospital
Other Study IDs: 670548
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-09

CONDITIONS: Distal Radius Fractures
Keywords: Wrist Fractures; Distal Forearm Fractures
MeSH Terms: conditions — Wrist Fractures | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a distal radius fracture: Dorsally displaced distal radius fractures reduced to an acceptable position in patients aged 18-65 years.
  Interventions: Radiation: X-ray (wrist)after 3 months and CT (wrist) the day after closed reduction

INTERVENTIONS:
Radiation: X-ray (wrist)after 3 months and CT (wrist) the day after closed reduction — One addition x-ray and on addition CT scan of the wrist

SUMMARY:
The study examines whether there are radiological criteria that can give an indication if a dorsally displaced distal radius fracture remains stable without the needs for surgery after closed reduction in patients between 18 and 65 years of age.

DETAILED DESCRIPTION:
1. Background

   Distal radius fracture is the most common fractures in adults, and there is agreement that there is a correlation between anatomical reduction and function in younger age groups (McQueen 1988, Cooney 1989). In the case of elderly patients (over 65 years), this is more debated (Egol 2010, Hassellund 2021, Panigrahi 2022).

   Dislocated distal radius fractures are initially treated with closed reduction and plaster (Arora 2011, Earnshaw 2002, Mackenney 2006). An unstable distal radius fracture is a fracture that dislocates after casting despite a successful reduction (Chung 2023). It is important to find out as early as possible whether a fracture is unstable only with a cast, so that these patients can be operated on without unnecessary delay, as a delayed operation can lead to reduced function (Selles 2021). Many have tried to come up with criteria that can predict whether the fracture is too unstable for plaster treatment only, but currently there are no standard criteria for this (Mackenney 2006, Lafontaine 1989, Nesbitt 2004, Abbaszadegan 1989, Tahririan 2013, Hove 1994, Leone 2004 ). Only increasing age, female gender and dorsal cortical comminution (all of which are factors that can indicate osteoporosis/osteopenia) have been shown to be significant criteria based on a meta-analysis from 2016 (Walenkamp 2016). However, there is a need for further studies of this, as practice now differs between the various hospitals in Norway, and also between different countries.

   According to the Norwegian guidelines, a distal radius fracture is considered for surgery based on certain radiological criteria. For patients under 65 years of age, it is strongly recommended to operate on a distal radius fracture if there is ≥ 10 degrees of dorsal angulation of the radius articular surface (from 90º on the longitudinal axis of the radius), ulnar variance ≥ 2 mm, intra-articular step ≥ 2 mm, incongruence in the distal radioulnar joint or cortical comminution in the fracture area/substance loss of the dorsal cortex of the distal radius before reduction. If one chooses conservative treatment for a well-reduced but possibly unstable fracture, it is good practice to follow the patient with regular X-ray checks. In American guidelines, there is a moderate recommendation to operate on fractures with dorsal tilt more than10 degrees, ulnar variance more than 3mm, intra-articular diastasis or step more than 2 mm after reduction. The recommendations behind the guidelines in Norway and in the USA are based on various studies with varying degrees of strength, as well as the surgeons experiences. Most of these studies include patients over 65 years of age, and increasing age has been shown to be one of the strongest indicators of whether a reduced fracture dislocates (Mackenney 2006). Many studies also exclude patients who have been set up directly for surgery without the criteria for why these patients have been considered for surgery being specified in more detail (Walenkamp 2016). Furthermore, most studies do not distinguish between displaced and minimally displaced fractures. Dorsal angulation that is accepted varies from 10-15 degrees from the neutral plane or 5 degrees from the starting point in various studies. Dorsal cortical comminution is not defined in most studies. Intra-articular fractures are often also included without any reflection on this. Some studies show that these are more unstable than extra-articular fractures (Lutz 2011). Although the meta-analysis (Walenkamp) from 2016 did not find that intra-articular fractures are more unstable, it was discussed whether part of the reason could be that many intra-articular fractures go straight to surgery and that only the least dislocated intra-articular fractures are considered for conservative treatment.
2. Problems and goal setting

   There is reason to ask whether the guidelines, especially the Norwegian ones, can lead to overtreatment, as clinical experience indicates that a portion of the distal radius fractures in patients between 18 and 65 years of age retain their position after closed reduction without surgery. In particular, this applies to extra-articular A fractures (based on the AO classification), as it has been shown that dorsal tilt is what most often triggers an indication for surgery (Cross 2022). Most people would agree that there is a difference between a comminuted, intra-articular fracture that is reduced to a suboptimal position, and a simple A2 fracture with a dorsal angulation of 20 degrees that is reduced to an anatomical position, but often this last group still ends up with surgery . There are no guidelines that separate these types of fractures. The question is how we can select the fractures that maintain their position after closed reduction. A closed reduction is considered successful when the most anatomical appearance of the bone is achieved. Whether the volar cortex is hooked on after reduction has been shown to be an important indication that a fracture holds its position (LaMartina 2015, Phillips 2014), but none of the guidelines in Norway, the USA, Great Britain or Denmark include this as a criterion. Only the Swedish guidelines have taken this into consideration. In addition, it should be considered whether patients between 50-65 years should be separated as a group, as many of these patients have osteoporosis/osteopenia.

   The following study is planned as part of the doctoral work of Ingrid Oftebro:

   Which radiological criteria can predict that the position of a distal radius fracture remains stable in the cast after closed reduction?

   Main quiestion:

   Can we find out which of the distal radius fractures maintain their position after closed reduction in patients between 18 and 65 years of age (with focus on volar hook and dorsal comminution)?

   It is important to find out whether some patients are unnecessary operated based on Norwegian and international guidelines. Needless operations can cause complications and stress for the patient that could have been avoided (Cross 2022, Rozental 2003). From a socio-economic perspective, it is also important to avoid unnecessary operations. Which radiological criteria before and after closed reduction of a distal radius fracture can help us to best predict whether a fracture retains its position in the cast?
3. Method

   The study is planned as a prospective study where consent will be obtained from the patient to look at various radiological criteria before and after reduction. Patients who are included must be between 18 and 65 years of age and have a dorsally displaced distal radius fracture that is reduced to an acceptable position (VLDV 75-95, RIV more than 15 degrees, ulnar variance less than 2 mm, step in the articular surface less than 2 mm) . Patients between 50-65 are more susceptible to osteoporosis/osteopenia, and we want to separate these as a group. All patients with low-energy fractures over the age of 50 are offered an osteoporosis examination at the OUS, and we can thus record the proportion of patients in this group who are diagnosed with osteoporosis/osteopenia.

   The patients will undergo normal closed repositioning with the traction method performed by LIS2 doctors/senior doctors and a plaster-technician/nurse. X-ray is taken before reduction, and X-ray and CT after reduction. X-ray will also be taken of the healthy side to be able to measure shortening more accurately, as there are anatomical variants.

   A common x-ray of the wrist consists of a PA projection (frontal projection) and a lateral projection with 15 degrees angulation (Medoff 2005).

   We will include extra-articular fractures (A2/3-fractures) and intra-articular fractures (C1/2-fractures) with intraarticulare step less than 2 mm before reduction.

   We want to examine the following radiological criteria (before and after repositioning): dorsal dislocation, ulnar variance, whether the volar cortex is hooked, to what extent there is a radial displacement/ad latus, radial inclination (RIV), radial height, dorsal, radial and ulnar comminution, carpal alignment and accompanying fracture of the ulna styloid process (avulsion fracture or at the base). In addition, we want to look at the extent to which the degree of dislocation before repositioning will affect whether the positions are maintained after repositioning.

   If a patient agrees to join the study, he or she will have a follow-up 6-8 days after reduction, where we will check if the fracture holds its position. If there is redislocation of the fracture beyond the limits mentioned above, the patient will be set up for surgery.

   X-rays before and X-rays and CT after reduction, as well as at follow-ups, will be examined with regard to the criteria mentioned above. Two experienced senior doctors at the out-patient clinic and a doctor specialising in orthopedic hand surgery at the orthopedic department OUS, Ullevål, will evaluate the X-rays, and where the measurements are not the same, the group will sit down to reach an agreement on the measurements. If the fracture has kept its position, they will be checked after another 6-8 days to check for late dislocation. If there is a slight redislocation within the above mentioned limits, a third follow-up will be scheduled within 3 weeks from injury. X-rays when the cast is removed (after 5 weeks) will also be examined in the patients where the fracture has maintained its position at the controls. The patients will take a final X-ray after 3 months.

   Complications such as CRPS (complex regional pain syndrome), osteotomy in the course due to symptomatic malunion, etc. will be recorded.

   We plan to include patients in a 2-year period from 01/10/2024 to 31/09/2026 at the outpatient clinic at the orthopedic department, OUS Ullevål (assumed N = 212). An experienced statistician from the University of Oslo will help with the calculations.
4. The importance of the project

The project will provide new knowledge about distal radius fractures in patients between 18 and 65 years of age and about the need for operative treatment after attempts at conservative treatment with closed reduction and casting. This knowledge will help to give the individual patient the best possible treatment so that unnecessary waiting for surgery and unnecessary operations are avoided. It will provide the opportunity to include new/more complementary criteria to the national guidelines in order to obtain better clinical assessment, and to avoid overtreatment. This will be important for the patients (avoid complications/burden by operating), as well as a socio-economic significance as surgery can lead to increased costs compared to conservative treatment with plaster. Distal radius fracture is the most frequently operated fracture in orthopedics, and there is therefore a large volume that can potentially be reduced.

ELIGIBILITY:
Inclusion criterias:

* 18-65 years old, living in Oslo/surroundings (available for follow-up)
* AO class A2/3 or C1/C2 fractures
* Dorsally displaced fracture of the distal radius (minimum VLDV more than100 or ulnar variance more than 2 mm compared to healthy side before reduction) with or without PSU fracture
* Reduced to an acceptable position (VLDV 75-95 degrees, RIV more than 15 degrees, ulnar variance more than 2 mm, step/diastasis in the joint surface less than 2 mm)

Exclution criterias:

* Volar comminution (AO A3.3), step/diastasis more than 2 mm before reduction
* Ad latus more than 2 cortex widths after reduction
* Bilateral fractures
* Open fractures
* Previous wrist fracture in adulthood
* Still open growth disc on X-ray
* Antebrachium or carpal fracture
* Ligament damage in the root of the hand or DRUJ
* Lack of compliance (dementia, psychiatry/drug abuse, etc.)
* Language problems
* Rheumatoid arthritis or other systemic disease that can affect the result

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the outpatient clinic at the Ortopedic department, Oslo University Hospital, Ullevål, with a dorsally displaced distal radius fracture, aged 18-65 years, reduced to an acceptable postition, included in a 2 year period (oct 2024 - oct 2026).
Sampling Method: Non-Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-10-07 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Radiological criterias 3 months after fracture | 3 months
  Whitch of the pre-defined radiological criterias (with a focus on dorsal comminution and volar hook) measured on x-ray before and after closed reduction can predict alignment 3 months after fracture

SECONDARY OUTCOMES:
CT criterias | 1 day after the fracture is reduced
  Grade different radiological criterias on CT, such as comminution and volar hook. Study intra/inter-observer reliability in these gradings.
How osteoporosis/osteopenia may affect instability in the age group 50-65 | 1 year
  Count how many of the patients aged 50-65 that have osteoporosis/osteopenia or who are assessed with this during the course of the study. (Assessment for osteoporosis/osteopenia is part of the ordinary clinical treatment program for patients over 50 years with a distal radius fracture.) Investigate whether those with osteoporosis/osteopenia have worse alignment on X-ray after 3 months than those without osteoporosis/osteopenia and whether the fractures in this age group have a greater tendency towards instability.

CONTACTS AND LOCATIONS:
Overall Officials: Lene B. Solberg, PhD MD, Principal Investigator — Division of Orthopaedic Surgery, Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Aker, Oslo Skadelegevakt, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No
The Norwegian law does not allow us to share IPD without a specific approval from the Regional Ethical Commitee (REC). If someone would like us to share IPD, we will consider to send an application to REC for this.

REFERENCES:
- [Background] McQueen M, Caspers J. Colles fracture: does the anatomical result affect the final function? J Bone Joint Surg Br. 1988 Aug;70(4):649-51. doi: 10.1302/0301-620X.70B4.3403617.
- [Background] Cooney WP. Management of Colles' fractures. J Hand Surg Br. 1989 May;14(2):137-9. doi: 10.1016/0266-7681_89_90112-5. No abstract available. PMID 2746109
- [Background] Egol KA, Walsh M, Romo-Cardoso S, Dorsky S, Paksima N. Distal radial fractures in the elderly: operative compared with nonoperative treatment. J Bone Joint Surg Am. 2010 Aug 4;92(9):1851-7. doi: 10.2106/JBJS.I.00968. PMID 20686059
- [Background] Hassellund SS, Williksen JH, Laane MM, Pripp A, Rosales CP, Karlsen O, Madsen JE, Frihagen F. Cast immobilization is non-inferior to volar locking plates in relation to QuickDASH after one year in patients aged 65 years and older: a randomized controlled trial of displaced distal radius fractures. Bone Joint J. 2021 Feb;103-B(2):247-255. doi: 10.1302/0301-620X.103B2.BJJ-2020-0192.R2. PMID 33517725
- [Background] Panigrahi TK, Ray S, Mallik M, Maharaj RC, Khatua J, Nanda DP. Determining the Borderline Anatomical Parameters for Better Functional Outcome of Colles Fracture: A Prospective Study. Rev Bras Ortop (Sao Paulo). 2021 May 5;57(4):619-628. doi: 10.1055/s-0041-1726062. eCollection 2022 Aug. PMID 35966419
- [Background] Arora R, Gabl M, Erhart S, Schmidle G, Dallapozza C, Lutz M. Aspects of current management of distal radius fractures in the elderly individuals. Geriatr Orthop Surg Rehabil. 2011 Sep;2(5-6):187-94. doi: 10.1177/2151458511426874. PMID 23569689
- [Background] Earnshaw SA, Aladin A, Surendran S, Moran CG. Closed reduction of colles fractures: comparison of manual manipulation and finger-trap traction: a prospective, randomized study. J Bone Joint Surg Am. 2002 Mar;84(3):354-8. doi: 10.2106/00004623-200203000-00004. PMID 11886903
- [Background] Mackenney PJ, McQueen MM, Elton R. Prediction of instability in distal radial fractures. J Bone Joint Surg Am. 2006 Sep;88(9):1944-51. doi: 10.2106/JBJS.D.02520. PMID 16951109
- [Background] Chung SR, Chung KC. Recognizing and Treating Unique Distal Radius Fracture Patterns that are Prone to Displacement. Hand Clin. 2023 Aug;39(3):279-293. doi: 10.1016/j.hcl.2023.02.004. Epub 2023 Mar 31. PMID 37453757
- [Background] Selles CA, Mulders MAM, Winkelhagen J, van Eerten PV, Goslings JC, Schep NWL; VIPAR Collaborators. Volar Plate Fixation Versus Cast Immobilization in Acceptably Reduced Intra-Articular Distal Radial Fractures: A Randomized Controlled Trial. J Bone Joint Surg Am. 2021 Nov 3;103(21):1963-1969. doi: 10.2106/JBJS.20.01344. PMID 34314402
- [Background] Lafontaine M, Hardy D, Delince P. Stability assessment of distal radius fractures. Injury. 1989 Jul;20(4):208-10. doi: 10.1016/0020-1383(89)90113-7. PMID 2592094
- [Background] Nesbitt KS, Failla JM, Les C. Assessment of instability factors in adult distal radius fractures. J Hand Surg Am. 2004 Nov;29(6):1128-38. doi: 10.1016/j.jhsa.2004.06.008. PMID 15576227
- [Background] Abbaszadegan H, Jonsson U, von Sivers K. Prediction of instability of Colles' fractures. Acta Orthop Scand. 1989 Dec;60(6):646-50. doi: 10.3109/17453678909149595. PMID 2624083
- [Background] Tahririan MA, Javdan M, Nouraei MH, Dehghani M. Evaluation of instability factors in distal radius fractures. J Res Med Sci. 2013 Oct;18(10):892-6. PMID 24497862
- [Background] Hove LM, Solheim E, Skjeie R, Sorensen FK. Prediction of secondary displacement in Colles' fracture. J Hand Surg Br. 1994 Dec;19(6):731-6. doi: 10.1016/0266-7681(94)90247-x. PMID 7706876
- [Background] Leone J, Bhandari M, Adili A, McKenzie S, Moro JK, Dunlop RB. Predictors of early and late instability following conservative treatment of extra-articular distal radius fractures. Arch Orthop Trauma Surg. 2004 Jan;124(1):38-41. doi: 10.1007/s00402-003-0597-6. Epub 2003 Nov 8. PMID 14608466
- [Background] Walenkamp MM, Aydin S, Mulders MA, Goslings JC, Schep NW. Predictors of unstable distal radius fractures: a systematic review and meta-analysis. J Hand Surg Eur Vol. 2016 Jun;41(5):501-15. doi: 10.1177/1753193415604795. Epub 2015 Sep 29. PMID 26420817
- [Background] Lutz M, Arora R, Krappinger D, Wambacher M, Rieger M, Pechlaner S. Arthritis predicting factors in distal intraarticular radius fractures. Arch Orthop Trauma Surg. 2011 Aug;131(8):1121-6. doi: 10.1007/s00402-010-1211-3. Epub 2010 Dec 15. PMID 21161253
- [Background] Cross GWV, Saini RS, Monem M, Sofat R. Analysis of Our Open Reduction and Internal Fixation of Distal Radius Fractures in Adults: Are We Over Operating? J Wrist Surg. 2021 Jul 2;11(1):48-53. doi: 10.1055/s-0041-1731384. eCollection 2022 Feb. PMID 35127264
- [Background] LaMartina J, Jawa A, Stucken C, Merlin G, Tornetta P 3rd. Predicting alignment after closed reduction and casting of distal radius fractures. J Hand Surg Am. 2015 May;40(5):934-9. doi: 10.1016/j.jhsa.2015.01.023. Epub 2015 Mar 12. PMID 25772286
- [Background] Phillips AR, Al-Shawi A. Restoration of the volar cortex: predicting instability after manipulation of distal radial fractures. Injury. 2014 Dec;45(12):1896-9. doi: 10.1016/j.injury.2014.09.007. PMID 25441173
- [Background] Rozental TD, Beredjiklian PK, Bozentka DJ. Functional outcome and complications following two types of dorsal plating for unstable fractures of the distal part of the radius. J Bone Joint Surg Am. 2003 Oct;85(10):1956-60. doi: 10.2106/00004623-200310000-00014. PMID 14563804
- [Background] Medoff RJ. Essential radiographic evaluation for distal radius fractures. Hand Clin. 2005 Aug;21(3):279-88. doi: 10.1016/j.hcl.2005.02.008. PMID 16039439
- [Background] Angst F, Aeschlimann A, Angst J. The minimal clinically important difference raised the significance of outcome effects above the statistical level, with methodological implications for future studies. J Clin Epidemiol. 2017 Feb;82:128-136. doi: 10.1016/j.jclinepi.2016.11.016. Epub 2016 Dec 14. PMID 27986610
- [Background] McCreary DL, Sandberg BC, Bohn DC, Parikh HR, Cunningham BP. Interpreting Patient-Reported Outcome Results: Is One Minimum Clinically Important Difference Really Enough? Hand (N Y). 2020 May;15(3):360-364. doi: 10.1177/1558944718812180. Epub 2018 Nov 21. PMID 30461316
- See also: Norwegian Guidelines for Distal Radius Fractures — https://files.magicapp.org/guideline/452ee86b-07d4-4e5e-9bb4-99fd6a26f5c8/2_6/pdf/published_guideline_549-2_6.pdf
- See also: British Guidelines for Distal Radius Fractures — https://www.bssh.ac.uk/_userfiles/pages/files/professionals/Radius/Blue%20Book%20DRF%20Final%20Document.pdf
- See also: Danish Guidelines for Distal Radius Fractures — https://www.sst.dk/da/udgivelser/2014/~/media/EB0328BE70DE4D4AB5C6E164EC87C3BA.ashx?m=.pdf
- See also: Swedish Guidelines for Distal Radius Fractures — https://d2flujgsl7escs.cloudfront.net/external/Nationellt+v%C3%A5rdprogram+f%C3%B6r+behandling+av+distala+radiusfrakturer.pdf